CLINICAL TRIAL: NCT03457987
Title: Preoperative Renal Functional Reserve to Predict Risk of Acute Kidney Injury After Cardiac Surgery: The IRRIV Task Force and Collaborators for the Prevention of Acute Kidney Injury
Brief Title: Acute Kidney Injury After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Shanghai Jiao Tong University School of Medicine (Other); Robert Bosch Medical Center (Other); Ospedale San Bortolo di Vicenza (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Faeq Husain-Syed, Senior Physician, University of Giessen
Other Study IDs: AZ 216/17
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-06

CONDITIONS: Acute Kidney Injury
Keywords: protein load; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators seek to determine whether a reduced preoperative renal functional reserve predicts postoperative acute kidney injury in patients with normal estimated glomerular filtration rates undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
Although acute kidney injury (AKI) frequently complicates cardiac surgery, methods to determine AKI risk in patients without underlying kidney disease are lacking. Renal functional reserve (RFR) can be used to measure the capacity of the kidney to increase glomerular filtration rate under conditions of physiological stress and may serve as a functional marker that assesses susceptibility to injury.

The investigators seek to determine whether a reduced preoperative RFR predicts postoperative AKI in patients with normal estimated glomerular filtration rates undergoing elective cardiac surgery. All centres will measure RFR with creatinine clearance, except University Hospital Giessen where in addition iohexol plasma-clearance will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 18 years
2. Subjects undergoing elective cardiac surgery (with or without cardiopulmonary bypass)
3. Subjects with an estimated GFR ≥60 ml/min/1.73 m2 (CKD-Epidemiology Collaboration equation)
4. Subjects who signed informed consent forms

Exclusion Criteria:

1. Preexisting acute kidney injury (as determined by all available serum creatinine values from hospital and outpatient medical records within the previous 90 days)
2. Chronic kidney disease ≥ stage III (KDIGO)
3. Subjects undergoing transcatheter aortic valve implantation (TAVI)
4. Pregnancy
5. Solitary kidney
6. Diabetes mellitus type 1
7. Recent cardiac arrest (within last 3 months)
8. Liver failure or cirrhosis
9. Total parenteral nutrition
10. Hemoglobin <11 g/dl
11. Sepsis
12. History of malabsorption, chronic inflammatory bowel disease, short bowel, or pancreatic insufficiency
13. Transplant donor or recipient
14. Active autoimmune disease with renal involvement
15. Rhabdomyolysis
16. Prostate hypertrophy with International Prostate Symptom Score ≥20
17. Active neoplasm
18. Decompensated heart failure / inability to pause angiotensin-converting enzyme inhibitors or angiotensin II receptor blockers minimum 2 days before protein load
19. Known iodine allergy (exclusion criteria only for those centres who use iohexol plasma clearance for determination of GFR)
20. TSH <0.3 µU/l (exclusion criteria only for those centres who use iohexol)
21. Subjects who received intravenous radiocontrast agents within the 72 hours before the protein load
22. Subjects who received NSAIDs within 48 hours before the protein load

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing elective cardiac surgery (with or without cardiopulmonary bypass) with an estimated GFR ≥60 ml/min/1.73 m2 (CKD-Epidemiology Collaboration equation)
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Whether a reduced preoperative RFR ≤15 ml/min/1.73 m2 increased the odds ratio for postoperative acute kidney injury in patients undergoing elective cardiac surgery. | Preoperative
  Renal functional reserve

SECONDARY OUTCOMES:
determine preoperative RFR accuracy based on receiver operating characteristic curve curve to predict acute kidney injury. | Preoperative
  Renal functional reserve
To analyze an acute kidney injury risk prediction model based on clinical covariates. | Preoperative
  Renal functional reserve
Mortality at 30 and 90 days | 30 and 90 days after surgery
  Mortality
Length of stay in intensive care unit and hospital. | Postoperative
  Hospital stay
Use and duration of renal replacement therapy during hospital stay. | Postoperative
  Renal replacement therapy
Renal replacement therapy dependence at days 30 and 90. | 30 and 90 days after surgery
  Renal replacement therapy
To evaluate renal function at three months after surgery. | 3 months after surgery
  Estimated glomerular filtration rate
To evaluate whether preoperative RFR is correlated to renal function at three months after surgery. | Preoperative
  Renal functional reserve
To evaluate whether chronic kidney disease is associated to preoperative RFR. | Preoperative
  Renal functional reserve

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, MD, Study Director — San Bortolo Hospital, Vicenza, Italy
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication.

REFERENCES:
- [Result] Husain-Syed F, Ferrari F, Sharma A, Danesi TH, Bezerra P, Lopez-Giacoman S, Samoni S, de Cal M, Corradi V, Virzi GM, De Rosa S, Mucino Bermejo MJ, Estremadoyro C, Villa G, Zaragoza JJ, Caprara C, Brocca A, Birk HW, Walmrath HD, Seeger W, Nalesso F, Zanella M, Brendolan A, Giavarina D, Salvador L, Bellomo R, Rosner MH, Kellum JA, Ronco C. Preoperative Renal Functional Reserve Predicts Risk of Acute Kidney Injury After Cardiac Operation. Ann Thorac Surg. 2018 Apr;105(4):1094-1101. doi: 10.1016/j.athoracsur.2017.12.034. Epub 2018 Jan 31. PMID 29382510
- [Result] Sharma A, Zaragoza JJ, Villa G, Ribeiro LC, Lu R, Sartori M, Faggiana E, de Cal M, Virzi GM, Corradi V, Brocca A, Husain-Syed F, Brendolan A, Ronco C. Optimizing a kidney stress test to evaluate renal functional reserve. Clin Nephrol. 2016 Jul;86(7):18-26. doi: 10.5414/CN108497. PMID 27285313
- [Result] Ronco C, Kellum JA, Haase M. Subclinical AKI is still AKI. Crit Care. 2012 Jun 21;16(3):313. doi: 10.1186/cc11240. PMID 22721504
- [Result] Husain-Syed F, Ferrari F, Sharma A, Hinna Danesi T, Bezerra P, Lopez-Giacoman S, Samoni S, de Cal M, Corradi V, Virzi GM, De Rosa S, Mucino Bermejo MJ, Estremadoyro C, Villa G, Zaragoza JJ, Caprara C, Brocca A, Birk HW, Walmrath HD, Seeger W, Nalesso F, Zanella M, Brendolan A, Giavarina D, Salvador L, Bellomo R, Rosner MH, Kellum JA, Ronco C. Persistent decrease of renal functional reserve in patients after cardiac surgery-associated acute kidney injury despite clinical recovery. Nephrol Dial Transplant. 2019 Feb 1;34(2):308-317. doi: 10.1093/ndt/gfy227. PMID 30053231